CLINICAL TRIAL: NCT06890975
Title: "F!reF!ghterF!t": A Randomized Controlled Trial of Lifestyle Coaching Interventions for Obese Firefighters
Brief Title: "F!reF!ghterF!t": Lifestyle Coaching Interventions for Obese Firefighters (FireFit)
Acronym: FireFit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Ardmore Institute of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHA-IRB-23-24-340
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: obesity; firefighters; diabetes mellitus; coaching; healthy lifestyle; lifestyle medicine; metabolic syndrome; quality of life; mental health; physical fitness
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Metabolic Syndrome; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Health Coaching versus written lifestyle instructions
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control/ General Written Health Instructions (No Intervention): Participants will receive standard lifestyle recommendations, consisting of two pages of written information summarized from the American Heart Association's 'Healthy for Good' webpages for the general public. These will include guidance on healthy diets, physical activity, healthy sleep, stress reduction, and avoiding tobacco, excess alcohol, and other harmful substances.
- Individual & Group Lifestyle Medicine-based Coaching (Active Comparator): This group will receive personal and group coaching sessions based on the six pillars of lifestyle medicine: 1) a plant- predominant eating pattern (consistent with the AIH "Full Plate Living" program); 2) physical movement; 3) restorative sleep; 4) management of stress; 5) avoidance of risky substances; and 6) positive social connections. Target goals for the participants assigned to Lifestyle Coaching will include the following: improving diet quality together with moderate caloric restriction; engaging in more physical activity with a goal of 150 minutes or more per week of at least moderate intensity (e.g. brisk walking); getting 7-8 hours of sleep nightly when possible and using short naps when work or other conditions interfere with getting at least 7 hours of sleep; increasing resilience and using positive social/family connections to manage/decrease stress.
  Interventions: Behavioral: Lifestyle Coaching

INTERVENTIONS:
Behavioral: Lifestyle Coaching — The schedule for the individual and group coaching sessions is summarized below:
  * Individual Coaching: Six one-on-one online sessions with a trained dietician, starting with an initial 30-minute session at baseline, followed by sessions at one month and then every other month.
  * Group Coaching: 60-minute group online sessions with up to 15 participants per group. Group sessions schedule: there will be a total of 13 group sessions. They will meet once a week for the first 4 weeks, twice monthly for the next 8 weeks of follow-up, and then monthly for the remaining follow-up until the 13th session.
  Arms: Individual & Group Lifestyle Medicine-based Coaching

SUMMARY:
Our goal is to explore the effectiveness of 9- month lifestyle medicine based coaching intervention (individual and group coaching) versus control (usual care/ written health instructions). The primary study outcomes will be mean changes in body composition metrics . Secondary outcomes will be the prevalence of metabolic abnormities, progression/regression of Metabolic Syndrome, push-up & sit/stand capacity, self-reported physical activity, and quality of life/diet/sleep measures.

DETAILED DESCRIPTION:
RATIONALE/GOALS: Obesity is a major health hazard in the US fire service. It contributes to excess cancer, cardiovascular disease and behavioral health issues. Obesity is negatively associated with 12/13 health priorities identified by the National Fallen Firefighter Foundation. Mitigating obesity is crucial to the fire service's goals of reducing chronic diseases and their adverse economic/operational impacts.

METHODS: At least 75 male firefighters self-reporting a body mass index (BMI) of >/= 30 kg/m2 AND interest in weight loss will complete a baseline health assessment including: lifestyle scores, body composition, metabolic/hormonal indices, physical fitness, and behavioral health screens, until 50 eligible firefighters have been consented and enrolled. After the initial clinical evaluation, 50 eligible firefighters will be randomized into the two study groups (about 25 firefighters to each arm): 1. General Health Instructions (CONTROL) and 2. Individual & Group Lifestyle Coaching based on the six pillars of Lifestyle Medicine & Full Plate Living. Participants will repeat the all health/fitness measures at 3-, 6- and 9-months post study entry. The two treatment groups will be compared on an intention to treat basis.

ANTICIPATED OUTCOMES: Compared to CONTROL, firefighters receiving the Lifestyle Coaching Intervention should achieve significantly greater improvements in body composition, metabolic & other health measures, as well as adopt healthy lifestyle behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Male firefighters aged 18-60 years
* Currently active as volunteer or career firefighters
* Body mass index (BMI) ≥30 kg/m² based on self-reported height and weight
* Express interest in participating in a clinical study aimed at improving body composition (weight loss), metabolic status, and quality of life
* Residing and/or working in Massachusetts, Rhode Island, or Southern New Hampshire (Boston metro area)

Exclusion Criteria:

* Female sex*
* BMI <30 kg/m² based on self-reported height and weight
* Active psychosis
* History or diagnosis (during the RCT) of any of the following:

Major cardiovascular disease event (e.g., myocardial infarction, cardiac arrest, cerebrovascular accident) Cancer (excluding non-melanoma skin cancer) Abnormal liver function (aminotransferase, bilirubin, or alkaline phosphatase ≥3× the upper limit of normal) Renal dysfunction (estimated glomerular filtration rate ≤30 mL/min/1.73 m²)

* Current or recent (within 6 months) use of testosterone treatment or anti-obesity/obesogenic medications
* Unwillingness to adhere to potential intervention assignments

  * Because this is an exploratory study, the number of subjects is limited, and men make up roughly 85% of the US fire service, the current proposal is limited to men. In future studies, we will include women firefighters.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in body mass index | From the start of the intervention to its conclusion at nine months.
  Body Mass Index (kg/m-squared)
Mean change in body fat | From the start of the intervention to its conclusion at nine months.
  Body fat percentage as measured by bioelectrical impedance
Mean change in waist circumference | From the start of the intervention to its conclusion at nine months.
  Waist circumference (cm)
Mean change in waist/hip ratio | From the start of the intervention to its conclusion at nine months.
  Waist/hip ratio (waist circumference (cm) divided by hip circumference (cm)

SECONDARY OUTCOMES:
Prevalence of Metabolic Syndrome | From the start of the intervention to its conclusion at nine months.
  Number (%) of participants with 3 or more metabolic syndrome components
Push-up capacity | From the start of the intervention to its conclusion at nine months.
  1-minute push-up capacity
Sit/stand capacity | From the start of the intervention to its conclusion at nine months.
  1-munute sit to stand completions
Self-reported Healthy Lifestyle Score | From the start of the intervention to its conclusion at nine months.
  Score based on self-reported health behaviors from a standardized survey tool with validated component metrics
Self-reported quality of life | From the start of the intervention to its conclusion at nine months.
  Score based on the validated Short Form-12 Health Survey (SF-12). The SF-12 generates two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS), each ranging from 0 to 100. Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge Health Alliance, Sommerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy concerns and data-use restrictions